CLINICAL TRIAL: NCT06944691
Title: Prevalence of Major Depressive Disorder in the Population of People Followed up for HIV PREP Consulting the Infectious Diseases Department of Saint-Antoine Hospital, APHP and in General Practices
Brief Title: Mental Health and PreP
Acronym: SAM-P
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: APHP241798
Record Dates: First submitted 2025-04-09; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Disorder in Patients Taking PrEP
Keywords: Depression; mental disorders; HIV; Pre-exposure Prophylaxis
MeSH Terms: conditions — Depression; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One group to study a prevalence (Other)
  Interventions: Other: Major depressive disorder scale

INTERVENTIONS:
Other: Major depressive disorder scale — Pass HDRS to patient taking PrEP to study prevalence of Major Depressive Disorder
  Other Names: Hamilton Depression Rating Scale (HDRS)

SUMMARY:
According to ANSM, by June 2023, almost 85,000 people living in France had initiated medical monitoring for HIV PrEP since 2016. Since 2021, HIV PrEP can be prescribed for the first time in community clinics, in addition to hospital structures such as CeGIDDs, or by doctors specialising in infectious diseases, making this preventive treatment for HIV more accessible. The population undergoing PrEP treatment is typically men who have sex with men (MSM), living in the Ile-De-France region, with an average age of 36 and social security cover.

In view of the growing number of people being monitored for HIV PrEP, particularly in general practice, which accounts for 80% of prescribers in private practice, and which will increase from 19% of initiations in 2021 to 42% in 2023, it seems essential not to ignore the occurrence of comorbidities, in order to better prevent or detect pathologies that may occur during the monitoring of these people. It appears that mental illnesses, and in particular major depressive disorder or anxiety disorders, as well as addictions, are present in many people receiving PrEP treatment. A study carried out in Canada found a prevalence of depressive disorders of almost 24%, alcohol use disorders for almost 32% and moderate to severe substance use for 43.3% of their study population. While some studies have highlighted the possibility of a reduction in anxiety, depression and addictions in patients using HIV PrEP, no study seems to have looked at the prevalence of depression in this specific population, which is exposed to more traumatic events, aggression or violence, and addictive behaviour, themselves associated with more depressive or anxious symptoms.

To date, there is little information on the psychiatric comorbidities of patients undergoing HIV PrEP, apart from elements purely associated with PrEP (compliance, adherence to treatment or follow-up). In the context of prevention as part of primary care monitoring, it seems necessary to better identify these comorbid pathologies in this specific population, using the opportunity of PrEP monitoring to initiate treatment where appropriate.

DETAILED DESCRIPTION:
Given the gradual opening up of general practitioners to the initial prescription and monitoring of PrEP, their role in the identification and prevention of mental illness remains more than useful, and they can compensate for certain shortcomings in the context of hospital monitoring, boasting a certain territorial proximity, greater availability and more comprehensive patient management. Given the lack of data in France on the prevalence of mental illness, and in particular of major depressive disorder, the investigator wanted to gain a better understanding of these psychiatric illnesses in our patients undergoing PrEP in general practices and hospitals, by carrying out questionnaires recommended by the Haute Autorité de Santé (HAS) for monitoring the general population. Our study will thus make it possible to improve the data concerning the prevalence of major depressive disorder in patients being monitored for PrEP, potentially playing a role in adherence to treatment. Secondly, this study aims to provide a better description of the risk factors for these mental pathologies in this specific population by describing socio-demographic characteristics and sexual behavior, and to determine whether or not PrEP takes precedence over psychiatric management and the prevalence of psychotropic drugs in patients undergoing PrEP treatment.

The investigator want to assess the prevalence of anxiety and depressive disorders using hetero-questionnaires recommended by the French National Authority for Health, namely the Hamilton Depression Rating Scale (HDRS) for depression. Our secondary aim is to investigate the potential clinical characteristics of these disorders in patients undergoing PrEP treatment, for future, more substantial studies. Thus, by carrying out these questionnaires, screening for these disorders could be accompanied by a change in their medical management, through standardized management of depression, as described by the HAS.

ELIGIBILITY:
Inclusion Criteria:

* Any adult being treated for HIV PrEP at one of the centres taking part in the study
* Have French social security coverage

Exclusion Criteria:

* Follow-up to HIV
* First consultation for PrEP
* Limited understanding of French to answer questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Major Depressive Disorder | at inclusion visit Day 1
  Pass questionnary to evaluate the prevalence of major depressive disorder

SECONDARY OUTCOMES:
Describe the factors associated with this psychiatric entity in the overall study population | at inclusion visit Day 1
  Pass questionary
Clinical characterization of depressive episodes | at inclusion visit Day 1
  Evaluate the contribution of questionary in the screening of depressive episodes with regard to the clinician's response
Description of the the treatment plan for depressive disorders, i.e. before or after PrEP monitoring | at inclusion visit Day 1
  Pass questionary
Prevalence of co-prescriptions | at inclusion visit Day 1
  Describe the prevalence of co-prescriptions of HIV PrEP and psychotropic drugs (drugs used to treat mental illness).

CONTACTS AND LOCATIONS:
Overall Officials: Thibault Chiarabini, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: No